CLINICAL TRIAL: NCT06879405
Title: The Effect of Labour Hopscotch Based Midwifery Care in Labor on Birth Outcomes, Labor Pain, Birth Comfort and Satisfaction: Randomized Controlled Study
Brief Title: The Effect of Labour Hopscotch Based Midwifery Care in Labor
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gamze Akpınar, midwife, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AtaturkU.
Record Dates: First submitted 2025-03-04; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Labor Hopscotch
Keywords: labor hopscotch; midwife; labor pain; birth satisfaction; midwifery care
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: The research is a randomized controlled experimental design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Experimental Group: Midwifery care based on labor hopscotch was applied. The midwife performed the practices in labor hopscotch step by step in the experimental group. The practices started when the dilation was 4-5 cm and each practice lasted 20 minutes. A 30-minute break was given between the practices. Visual posters showing the practice steps were hung in the delivery rooms. According to the visual poster, the pregnant woman approaches the baby's footprint with each step she takes, and this situation increases the pregnant woman's motivation while ensuring her active participation in the practices. In women who experienced discomfort during the practices, the practices were paused for 10-15 minutes and then tried again. In case of discomfort again, the practices were not continued and the pregnant woman was removed from the study group.
  Interventions: Other: The Labor Hopscotch
- control group (No Intervention): Control Group: Pregnant women in this group continued to receive routine delivery room midwifery care in accordance with the concept of a mother-friendly hospital. Pregnant women give birth with minimal intervention and invasive procedures. If deemed necessary by the physician, interventions such as induction, propess, amniotomy, forceps/vacuum can be performed. NST is evaluated once an hour and vaginal examination is performed once every 2 hours (durations may vary according to the physician's request). If the pregnant woman wishes, labor can be monitored with a companion of her choice. Unless otherwise indicated, oral intake of pregnant women is not restricted.

INTERVENTIONS:
Other: The Labor Hopscotch — Labor Hopscotch consists of 4 basic parameters including movement (mobilization), positioning (birth stool, sitting on the toilet, birth ball, birth mat), water therapy and non-pharmacological methods for reducing pain. There are sub-contents for each of these parameters and hopscotch consists of 7 steps in total. Labor Hopscotch Model Steps;
  Step 1: Mobilization (squat, pelvic tilt, using stairs, movement) Step 2: Birth Stool (oral fluid support, massage, breathing techniques) Step 3: Sitting on the Toilet (urinating, dim lighting, music) Step 4: Water Therapy (Warm shower, breathing techniques, Squat, oral fluid support) Step 5: Birth Ball (drawing 8 with the birth ball, slow movement techniques) Step 6: Birth Mat (massage, exercise on the mat, quadruped position) Step 7: Alternative Methods (massage, aromatherapy).
  Arms: Experimental Group

SUMMARY:
This study aimed to evaluate the effects of labor hopscotch midwifery care on birth outcomes, labor pain, birth comfort and satisfaction. The research is a randomized controlled experimental design. The study will be conducted between June 1, 2024 and December 1, 2025 at the Tuzla State Hospital Maternity Unit affiliated with the Istanbul Provincial Health Directorate. The universe of the study consists of primiparous pregnant women who applied to the relevant maternity ward. A priori power analysis was used to determine the sample size of the study. The sample size was determined using the G*Power program version 3.1.9.7 (Heinrich-Heini-Universitat-Düsseldorf, Germany) and Cohen's standard effect sizes were used as a reference method in the power analysis. The sample size was calculated as 84 pregnant women (Experimental group: 42 pregnant women, Control group: 42 pregnant women). It was decided to collect data from a total of 100 pregnant women by including a 20% spare sample in case of data loss. For randomization, columns between 1-100 were created in the system using the Random Integer Generator method under the Numbers subheading of the random.org website. Considering the numbers 1 and 2 in the column, pregnant women who came to the delivery room were randomly assigned to these numbers (https://www.random.org/). Which number constituted which group was determined by drawing lots at the beginning of the study, and the result of the drawing was determined as 1 control group and 2 experimental groups. Experimental and control group data were collected simultaneously. In collecting the data, the Introductory Information Form, Birth Outcomes Form, Perineal Laceration Assessment Form, Visual Analog Scale (VAS), Birth Comfort Scale and Birth Satisfaction Scale Revised Form were used. In collecting the data, the Introductory Information Form, Birth Outcomes Form, Perineal Laceration Assessment Form, Visual Analog Scale (VAS), Birth Comfort Scale and Birth Satisfaction Scale Revised Form were used.

DETAILED DESCRIPTION:
Experimental Group: Midwifery care based on labor hopscotch was applied. The midwife performed the practices in labor hopscotch step by step in the experimental group. The practices started when the dilation was 4-5 cm and each practice lasted 20 minutes. A 30-minute break was given between the practices. Visual posters showing the practice steps were hung in the delivery rooms. According to the visual poster, the pregnant woman approaches the baby's footprint with each step she takes, and this situation increases the pregnant woman's motivation while ensuring her active participation in the practices. In women who experienced discomfort during the practices, the practices were paused for 10-15 minutes and then tried again. In case of discomfort again, the practices were not continued and the pregnant woman was removed from the study group.

Labor Hopscotch consists of 4 basic parameters including movement (mobilization), positioning (birth stool, sitting on the toilet, birth ball, birth mat), water therapy and non-pharmacological methods for reducing pain. There are sub-contents for each of these parameters and hopscotch consists of 7 steps in total. Labor Hopscotch Model Steps;

Step 1: Mobilization (squat, pelvic tilt, using stairs, movement) Step 2: Birth Stool (oral fluid support, massage, breathing techniques) Step 3: Sitting on the Toilet (urinating, dim lighting, music) Step 4: Water Therapy (Warm shower, breathing techniques, Squat, oral fluid support) Step 5: Birth Ball (drawing 8 with the birth ball, slow movement techniques) Step 6: Birth Mat (massage, exercise on the mat, quadruped position) Step 7: Alternative Methods (massage, aromatherapy).

Control Group: Pregnant women in this group continued to receive routine delivery room midwifery care in accordance with the concept of a mother-friendly hospital. Pregnant women give birth with minimal intervention and invasive procedures. If deemed necessary by the physician, interventions such as induction, propess, amniotomy, forceps/vacuum can be performed. NST is evaluated once an hour and vaginal examination is performed once every 2 hours (durations may vary according to the physician's request). If the pregnant woman wishes, labor can be monitored with a companion of her choice. Unless otherwise indicated, oral intake of pregnant women is not restricted.

Both experimental and control groups; In labor follow-up; Birth outcomes form was applied. In the experimental group, VAS application was applied after each of the 7 application steps in the labor hopscotch application and when the cervical dilatation was 4-5 cm, 8 cm, 10 cm. In the control group, VAS application was applied when the cervical dilatation was 4-5 cm, 8 cm, 10 cm. Birth Comfort Scale was applied to the pregnant women in the experimental and control groups when the cervical dilatation was 8-10 cm.

In the second stage of labor; Birth outcomes form and VAS application were applied to the pregnant women in both groups.

In the 3rd stage of labor; perineal laceration form was used for evaluation of the pregnant women in both groups.

Within the first 2 hours after birth; VAS and Birth Satisfaction Scale Revised Form were applied to the pregnant women in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Being literate
* Being between 18-45 years old
* Primigravida
* Having a single fetus
* Cervical dilatation of at most 4-5 cm
* Being open to communication
* Voluntarily participating in the study

Exclusion Criteria:

* Being over 45 years
* Multiparity
* High-risk pregnancy
* Progressing labor
* Having a diagnosed psychiatric illness

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 18 and over, pregnant women
Enrollment: 100 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | VAS will be applied during labor (after active phase).
  VAS is used to measure perceived pain. The scale has numbers from 1 to 10 on a vertical line. Number 1 symbolize almost none and number 10 symbolizes severe pain.
Birth Outcomes Form | Birth outcomes form will apply immediately after birth (second stage of labor).
  The form includes 13 questions that evaluate the duration of labor stages, interventions used during labor (induction, amniotomy, propess application, vacuum/forceps, other situations), data regarding the newborn (gender, height, weight, APGAR score, oxygen saturation, complication status, special care status), and satisfaction with the birth control application steps.
Perineal Laceration Evaluation Form | Perineal laceration form will be apply immediately delivery of the placenta (In the 3rd stage of labor).
  The form is a form created to evaluate postpartum episiotomy, perineal and cervical laceration status.
Birth Comfort Scale | Birth Comfort Scale will be apply before the baby is born.
  The scale consists of 9 items and 3 sub-dimensions (physical, psychospiritual and environmental). Each item is expected to be answered considering the comfort in the delivery room. Each item in the scale is scored between 1-5 (1=Strongly disagree, 2=Mostly disagree, 3=Partially agree, 4=Mostly agree, 5=Totally agree). The minimum score that can be obtained from the scale is 9, and the maximum score is 45. As the score increases, it indicates a high level of comfort, and as it decreases, it indicates a low level of comfort.
Birth Satisfaction Scale Revised Form | Birth Satisfaction Scale Revised Form will be apply within the first 2 hours after birth.
  It is a measurement tool consisting of 10 items and 3 sub-dimensions, applied to women who gave birth normally in the first ten days postpartum.6 items on the scale are positive, 4 items are negative, and 4 items are reverse scored. As the score on the scale increases, the woman's birth satisfaction increases.Birth Satisfaction Scale Revised Form will be apply to the pregnant women in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ayla Kanbur, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University, Erzurum, yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No